CLINICAL TRIAL: NCT06424899
Title: A Randomized, Controlled, Multicenter Phase II Clinical Study Comparing Neoadjuvant Chemoimmunotherapy and Immuno-consolidationafter Compared With Immunoconsolidation After Radical Chemoradiotherapy for Stage III Potentially Resectable NSCLC
Brief Title: A Study Comparing Neoadjuvant Chemoimmunotherapy and Immuno-consolidationafter Compared With Immunoconsolidation After Radical Chemoradiotherapy for Stage III Potentially Resectable NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zeng Jian (Other)
Responsible Party: Sponsor-Investigator, Zeng Jian, Archiater, Thoracic Surgery Department, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2024-106
Record Dates: First submitted 2024-05-10; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Platinum Compounds

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant: adebrelimab combined with platinum-based chemotherapy (Experimental): Adebrelimab 20mg/kg combined with platinum-based chemotherapy, q3w, MDT after 3 cycles, if the patient is suitable for surgery, surgery will be performed, and Adebrelimab adjuvant therapy will be performed for 35 cycles after surgery or until the disease recurrence or toxicity is difficult to tolerate as indicated by imaging; If the patient is not eligible for surgery after evaluation,, radical chemoradiotherapy will be performed, followed by Adebrelimab consolidation therapy for 35 cycles or until radiographically indicated disease recurrence or toxicity is difficult to tolerate.
  Interventions: Drug: Adebrelimab; Radiation: radical chemoradiotherapy; Drug: Platinum based chemotherapy
- radical chemoradiotherapy and adebrelimab consolidation for 38 cycles (Active Comparator): Consolidation therapy with adebrelimab , 20mg/kg, q3w, d1, was started within 1 to 42 days after radical chemoradiotherapy. The infusion time of adebrelimab was 60 minutes or more, and the treatment lasted for 38 consecutive cycles or until the disease recurred or the toxic reaction was difficult to tolerate as indicated by imaging.
  Interventions: Drug: Adebrelimab; Radiation: radical chemoradiotherapy; Drug: Platinum based chemotherapy

INTERVENTIONS:
Drug: Adebrelimab — This product is administered by intravenously guttae. The recommended dose of subcutaneous injection is 20mg/kg, administered every 3 Weeks (Q3W).
  Other Names: SHR-1316
Radiation: radical chemoradiotherapy — The total dose of radiotherapy was 60 Gy ± 10% (54 Gy - 66 Gy). The minimum technical standard for radiotherapy is the three dimensional conformal radiotherapy (3D-CRT) planned by CT.
Drug: Platinum based chemotherapy — Platinum based chemotherapy: Platinum drug must be one of cisplatin, carboplatin or nedaplatin; The other drug must contain one of the following: etoposide, vinorelbine, vinblastine, pemetrexed, taxanes (e.g., paclitaxel, docetaxel, albumin paclitaxel, paclitaxel liposomes) or gemcitabine (gemcitabine is not permitted in concurrent chemoradiotherapy regimens).

SUMMARY:
To evaluate the efficacy and safety adebrelimab in Combination with chemotherapy after 3 cycles as neoadjuvant therapy and surgery or chemoradiotherapy based on MDT compared with adebrelimab after chemoradiotherapy in potentially operable stage III NSCLC.

DETAILED DESCRIPTION:
In recent years, tumor immunotherapy has become an important means of clinical treatment of tumor. The emergence of immunotherapy has provided a new direction for the exploration of neoadjuvant therapy for non-small cell lung cancer. The purpose of this study is to compare the use of adebrelimab in patients with stage III potentially resectable locally advanced NSCLC (non-small cell lung cancer). The study will directly compare the curative chemoradiotherapy plus immune maintenance therapy model (Pacific model) with the neoadjuvant immune therapy plus curative surgery plus immune maintenance therapy model (Keynote-671 model). This comparison aims to provide a basis for determining treatment plans for patients with locally advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years old;
* 2. Histologically or cytologically confirmed non-small cell lung cancer. If the pathological type of the patient is adenocarcinoma, genetic testing should be performed to exclude EGFR/ALK mutations. Tumor tissue should be the first choice for genetic testing. If sufficient tumor tissue is not available, genetic testing using serum can be performed.
* 3. According to AJCC 8th Edition, the patient had stage IIIA-IIIB (T1-4N2M0). N2 was a non-giant type with lymph node diameter ≤3cm and no invasion or exocapsular invasion. Pathological biopsy of mediastinal lymph nodes is recommended to be clear, and patients without pathology should at least meet the short diameter of enhanced chest CT ≥1cm and high metabolism of PET-CT.
* 4. All lesions (including primary lesions and lymph nodes/metastases evaluated as metastases) of the patient should be evaluated jointly by surgeons, radiologists, and radiologists to be potentially resectable.
* 5. Subjects must have measurable target lesions (according to RECIST 1.1 criteria);
* 6. ECOG behavior status score 0-1;
* 7. No previous history of other malignant tumors;
* 8. Never received anti-tumor therapy such as surgery, radiotherapy, chemotherapy, targeted therapy and immunotherapy related to non-small cell lung cancer;
* 9. The patient should have adequate cardiopulmonary function: FEV1 and DLCO of the patient were ≥50% of the predicted value, and the ultrasonography suggested LVEF≥55%, and no clear signs of heart failure and severe coronary artery stenosis were found in various tests. The cardiopulmonary function was assessed by the surgeon as being able to tolerate surgical treatment.
* 10.The functional level of all vital organs must meet the following requirements:

  1. Bone marrow: absolute neutrophil count (ANC) ≥1.5× 109/L, platelet ≥100 × 109/L, hemoglobin ≥9 g /dl;
  2. Good coagulation function: defined as International standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
  3. Liver: total bilirubin ≤1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5 times the upper limit of normal;
  4. Kidney: serum creatinine ≤1.25 times the upper limit of normal or creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min;
* 11. Fertile men and women of childbearing age must consent to effective contraceptive use from the time they sign the master informed consent until 180 days after the final administration of the study drug. Women of reproductive age include premenopausal women and women within 2 years after menopause. Pregnancy test results of women of reproductive age must be negative within ≤ 7 days before the first study drug administration;
* 12. Voluntary participation in clinical research; Fully understand and know this study and sign ICF (Informed Consent).

Exclusion Criteria:

* 1. All lesions could not be completely resected by surgery;
* 2. Have any active autoimmune disease or history of autoimmune disease (such as uveitis, enteritis, hepatitis, pituitaritis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (may be included after hormone replacement therapy), tuberculosis); Patients with complete remission of childhood asthma without any intervention or vitiligo in adulthood could be included, but patients requiring medical intervention with bronchodilators could not be included;
* 3. Have a congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (HCV antibody positive and HCV-RNA above the lower detection limit of analytical methods), or co-infection with hepatitis B and hepatitis C;
* 4. There is a third lacunar effusion that is difficult to control, such as a large amount of pleural effusion or ascites or pericardial effusion;
* 5. Subjects requiring systemic therapy with corticosteroids (>10 mg/ day of prednisone or equivalent) or other immunosuppressants within 14 days prior to initial medication. In the absence of active autoimmune disease, inhaled or topical corticosteroids are permitted, as well as adrenal hormone replacement therapy at doses > 10 mg/ day of prednisone efficacy;
* 6. Subjects who have been treated with anti-tumor vaccine or other immunostimulating anti-tumor drugs (interferon, interleukin, thymosin, immunocell therapy, etc.) within 1 month before the first administration;
* 7. Participants who are participating in another clinical study or whose first dose is less than 4 weeks (or 5 half-lives of the investigational drug) since the end (last dose) of the previous clinical study;
* 8. Evidence of past or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiological pneumonia, drug-induced pneumonia, and severe impairment of lung function;
* 9. Major surgery, open biopsy, or significant trauma were performed within 28 days prior to enrollment;
* 10. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* 11. Pregnant or lactating women; A fertile patient who is unwilling or unable to take effective contraceptive measures;
* 12. Known allergic reactions, hypersensitivities, or intolerances to study drugs;
* 13. There are other circumstances in which the investigator considers it inappropriate to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-05-19 (Estimated); Primary Completion 2027-05-19 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
2 year EFS rate | Up to 2 years
  From the start of randomization to 2 years, the proportion of participants who experience any of the following events: disease progression making surgical treatment impossible, local or distant recurrence, or death due to any cause.
  Event-free Survival (EFS) is a term commonly used in the context of clinical trials and oncology to describe a period during which a patient with a disease, typically a cancer, remains free from any adverse events that are of clinical significance.

SECONDARY OUTCOMES:
OS | Up to 2 years
  Overall Survival, the time from the date of randomization until the death of the participant or the last follow-up.
TTDM | Up to 2 years
  the time from the initial diagnosis of a cancer until the first occurrence of distant metastasis.
TRAEs | Up to 2 years
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No